CLINICAL TRIAL: NCT04051008
Title: CTSI Pilot: Improving Adherence to a Diabetic Diet With a Grocery Shopping Intervention
Brief Title: CTSI Pilot: Improving Adherence to Diabetic Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Stephanie Anzman-Frasca, Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003054; UL1TR001412 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-09 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2; Diet, Healthy; Pre-diabetes
Keywords: grocery shopping; online shopping; diabetes; behavioral economics; diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Control (No Intervention): No intervention - participants will shop in-person as they usually would. Participants will receive recipe cards that follow the evidence-based DASH diet and correspond to dietary recommendations for diabetic patients.
- Group 2 - Online (Experimental): Participants will utilize online grocery shopping (shopping at a local grocery store via an online platform). Participants will also receive recipe cards that follow the evidence-based DASH diet and correspond to dietary recommendations for diabetic patients.
  Interventions: Behavioral: Online - use of online grocery shopping platform
- Group 3 - Default (Experimental): The default intervention will augment the Online intervention, showing participants a default cart when they log into their online grocery shopping accounts. They will be told that their cart has been filled with items that conform to a diabetic diet and can be used to make recipes from the provided recipe cards, and that they can modify it as they like. Participants will also receive recipe cards that follow the evidence-based DASH diet and correspond to dietary recommendations for diabetic patients.
  Interventions: Behavioral: Default - use of online grocery shopping platform with default shopping carts

INTERVENTIONS:
Behavioral: Online - use of online grocery shopping platform — The Online intervention will utilize online grocery shopping (shopping at a local grocery store via online platform).
  Arms: Group 2 - Online
Behavioral: Default - use of online grocery shopping platform with default shopping carts — The Defaults intervention, will augment the Online intervention, showing participants a default cart when they log into their online grocery shopping accounts. They will be told that their cart has been filled with items that conform to a diabetic diet and can be used to make the recipes from provided recipe cards, and that they may modify their cart as they like.
  Arms: Group 3 - Default

SUMMARY:
425 million adults live with diabetes worldwide, and the prevalence of Type 2 diabetes is rising. Dietary approaches are recommended for weight control and diabetes management, but modern environments, characterized by plentiful, unhealthy foods, pose challenges to selecting a healthy diet. Behavioral economics offers a framework for modifying the food environment to encourage individuals with diabetes to select low-calorie and low-sugar foods. The goal of this study is to test novel approaches informed by behavioral economics to promote healthier grocery shopping among diabetic patients. Adults who have Type 2 diabetes or who are at risk for developing Type 2 diabetes will be recruited. Participants will be randomly assigned to 1 of 2 interventions or a control group in which they will shop in-person as usual. The Online intervention will utilize online grocery shopping to promote healthier purchasing. The Defaults intervention will augment this intervention, showing participants a default shopping cart pre-filled with items that correspond to the DASH diet and diabetic diet goals, which they may modify as they like. Receipt data will be collected to quantify the alignment of purchases with diabetic diet goals before, during, and after interventions. Purchases lower in calories, carbohydrates, and sugar and higher in nutritional quality (DASH diet score) are expected in the Defaults group; the Online group is expected to have intermediary results between Defaults and Controls. The investigators will also explore effects of the interventions on spending and dietary intake. This study is intended to demonstrate the efficacy of strategies that leverage behavioral economics principles to make the purchasing of healthier foods easier. The strategies have translational significance as they could be incorporated into clinical treatment, with the potential to improve dietary intake, glucose regulation, weight, and medication needs among diabetic patients.

DETAILED DESCRIPTION:
The goal of this study is to test the effects of interventions informed by behavioral economics on the healthfulness of grocery purchases among diabetic adults. This study has a 3-group experimental design; adult patients with diabetes or at risk for diabetes who typically grocery shop in-person will be randomly assigned to one of two interventions or a control group. In all groups, recipe cards that follow the evidence-based DASH diet and correspond to dietary recommendations for diabetic patients will be provided. In addition, the first intervention, Online, will utilize online grocery shopping at a local grocery store to promote healthier purchasing, with a goal of removing visceral factors that can lead to impulse purchases in stores. The second intervention, Defaults, will augment the Online intervention, showing participants a default shopping cart when they log into their accounts. They will be told that their cart has been filled with items that conform to a diabetic diet and can be used to make the recipes from the provided recipe cards, and that they may modify their carts as they like. In the control group, participants will shop in-person as usual.

At baseline, all participants will complete a survey online or via phone and then will grocery shop in-person as usual. Participants will then be randomized and receive further instructions. For the next 3 weeks, they will receive recipe cards and shop in accordance with their assigned study group. The following week (post), they will grocery shop using the mode of their choice (in-person or online) and complete a survey again. Household receipt data will be collected throughout the study. The baseline period will also serve as a run-in period, and participants whose diabetes/prediabetes status is not confirmed by a physician or who do not comply with study guidelines for baseline procedures will not be randomized for further participation. Primary analyses will examine intervention effects on grocery purchases, with additional analyses examining spending and dietary intake. All participant interactions will occur online or via phone, with cards for participant payment sent via postal mail.

The specific aims of this study are: (1) to test effects of Online and Defaults interventions on diabetic adults' grocery purchases and (2) to explore effects of the Online and Defaults interventions on participants' spending during grocery shopping. It is hypothesized that (1a) purchases made by adults in the Defaults group will be lower in calories, carbohydrates, and sugar and higher in nutritional quality (DASH diet score) at post-test versus other study groups, (1b) adults in the Defaults group will show the greatest increases in nutritional quality versus other study groups, (1c) the Online group will have intermediary results between Defaults and Controls, and (2) there will be no difference in total dollars depicted on receipts across study groups during the intervention period (i.e. the costs of online shopping will be offset by effects of the Online and Default interventions).

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old
* Must have been diagnosed diabetes or demonstrate diabetes risk as defined by the American Diabetes Association
* Must shop in-person at select local grocery stores at least weekly, and at least 75% of the grocery shopping for the household must be done at these stores
* Must do at least 75% of the grocery shopping for the household
* Must speak English

Exclusion Criteria:

* Is under 18 years of age
* Does not meet diabetes/risk for diabetes criteria
* Does not shop in-person at select local grocery stores at least weekly
* Does not live in a household in which 75% of groceries come from select local grocery stores
* Does not do at least 75% of the grocery shopping for the household
* Does not speak English
* Receives SNAP or WIC benefits (an exclusion criterion for this study due to incompatibility of EBT cards with the selected online grocery shopping platform at this time)
* Has dietary restrictions or preferences that would not allow them to reasonably partake in the study (i.e. they would not be willing or able to buy/eat many of the staple foods included in default carts/recipe cards)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Anzman Frasca, PhD, Principal Investigator — Associate Professor
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hollis-Hansen K, Tan S, Bargnesi S, McGovern L, Drozdowsky J, Epstein LH, Leone LA, Mak E, Masci J, Anzman-Frasca S. Feasibility and implementation of a grocery shopping intervention for adults diagnosed with or at-risk for type 2 diabetes. Public Health Nutr. 2023 Oct;26(10):2118-2129. doi: 10.1017/S1368980023001453. Epub 2023 Jul 27. PMID 37496394

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Started | 21 | 21 | 23
Completed | 19 | 21 | 22
Not Completed | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The sample size for the baseline analysis population is different from the Participant Flow information because 1 participant did not have usable baseline survey data. Therefore there are n=64 baseline participants included in this section and n=65 randomized participants overall.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default | Total
Number analyzed (Participants) | 20 | 21 | 23 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (9.3) | 49.2 (12.8) | 53.7 (8.8) | 53.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 19 | 54
  Male | 3 | 3 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 20 | 22 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 19 | 18 | 21 | 58
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 23 | 64
Education [Count of Participants; unit: Participants]
  High school graduate or equivalent | 1 | 0 | 1 | 2
  Some college/associate's degree | 5 | 6 | 6 | 17
  Bachelor's degree | 6 | 5 | 8 | 19
  Graduate degree | 8 | 10 | 8 | 26
Total energy purchased [Mean (Standard Deviation); unit: kcal] | 26116.3 (26229.4) | 25832.2 (26229.4) | 25481.3 (16266.5) | 25799.8 (21272.6)
Total carbohydrates purchased [Mean (Standard Deviation); unit: grams] | 3335.7 (3175.3) | 2944.1 (2886.1) | 3009.2 (2269.0) | 3093.7 (2748.2)
Total sugar purchased [Mean (Standard Deviation); unit: grams] | 1289.7 (1243.9) | 1355.7 (1132.9) | 1345.5 (1065.4) | 1330.8 (1129.4)
Nutritional quality of grocery purchases [Mean (Standard Deviation); unit: units on a scale] — Nutritional quality of grocery purchases was created using indicators adapted from Fung 2008: fruit, vegetables, nuts/legumes, whole grains, low-fat dairy, sodium, red/processed meat, carbohydrates. Quintiles were calculated for each, using the number of items from a food group or sodium [mg] and carbohydrates [g] purchased that week. Resulting scores from 1-5 indicate whether participants were lower or higher on each indicator (red meat, sodium, carbohydrates reverse scored). The 8 scores were summed for a total nutritional quality score ranging from 8 to 40 (40=highest nutritional quality).
  units on a scale | 22.4 (4.5) | 22.4 (3.5) | 22.9 (4.8) | 22.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Calories Purchased
Description: Receipt data will be entered into Nutritionist Pro software and will be used to calculate total calories purchased from target grocery stores.
Time Frame: At post-test (week 5)
Population: The sample sizes reflect the number of participants in each group who provided receipt data during Week 5 of the study
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
Kcal | 24443.30 (14918.22) | 25339.20 (19069.60) | 18527.35 (15025.35)

2. Primary Outcome: Calories Purchased
Description: Receipt data are entered into Nutritionist Pro software and used to calculate total calories purchased from target grocery stores each week. For this analysis, the weekly values were aggregated, such that the least squares means reported herein represent average calories purchased across all 5 weeks, in the context of the repeated measures ANOVA model.
Time Frame: Weeks 1-5 (testing overall main effect of study group)
Population: All randomized participants were included in the repeated measures ANOVAs assessing the overall main effect of study group. Means reported below are least squares means representing calories purchased in each group overall across the time points
Measure: Least Squares Mean (Standard Deviation); unit: Kcal
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 21 | 21 | 23
Kcal | 25768 (14908.1) | 23479 (14870.5) | 20236 (14948.3)

3. Primary Outcome: Change in Calories Purchased
Description: Receipt data will be entered into Nutritionist Pro and will be used to calculate changes in total calories purchased from target grocery stores.
Time Frame: Baseline (week 1), intervention (weeks 2-4), and post-test (week 5)
Population: The intent of this analysis was to examine whether there were group differences in change in the specified outcome among all participants randomized. We report here the difference in least squares means within each group from week 1 to week 5.
Measure: Least Squares Mean (Standard Error); unit: kilocalories
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
kilocalories | -2661.91 (4023.56) | -1533.34 (4016.82) | -6892.76 (3786.38)

4. Primary Outcome: Carbohydrates Purchased
Description: Receipt data will be entered into Nutritionist Pro and will be used to calculate carbohydrates purchased from target grocery stores.
Time Frame: At post-test (week 5)
Population: Represents those with receipt data at post-test (week 5)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
grams | 3320.09 (2231.52) | 3153.88 (2805.51) | 2417.95 (2056.82)

5. Primary Outcome: Carbohydrates Purchased
Description: Receipt data are entered into Nutritionist Pro and used to calculate carbohydrates purchased from target grocery stores each week. For this analysis, the weekly values were aggregated, such that the least squares means reported herein represent average carbohydrates (grams) purchased across all 5 weeks, in the context of the repeated measures ANOVA model.
Time Frame: Weeks 1-5 (testing overall main effect of study group)
Population: All randomized participants were included in the repeated measures ANOVAs assessing the overall main effect of study group. Means reported below are least squares means representing carbohydrates purchased in each group overall across the time points
Measure: Least Squares Mean (Standard Deviation); unit: grams
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 21 | 21 | 23
grams | 3200.85 (1961.80) | 2760.89 (1955.66) | 2502.41 (1968.88)

6. Primary Outcome: Change in Carbohydrates Purchased
Description: Receipt data will be entered into Nutritionist Pro and will be used to calculate changes in carbohydrates purchased from target grocery stores.
Time Frame: Baseline (week 1), intervention (weeks 2-4), and post-test (week 5)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
grams | -102.78 (621.18) | -119.84 (620.36) | -575.67 (588.96)

7. Primary Outcome: Sugars Purchased
Description: Receipt data will be entered into Nutritionist Pro and will be used to calculate sugars purchased from target grocery stores.
Time Frame: At post-test (week 5)
Population: Represents those with receipt data at post-test (week 5)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
grams | 1212.27 (985.07) | 1026.31 (809.66) | 1024.99 (873.16)

8. Primary Outcome: Sugars Purchased
Description: Receipt data are entered into Nutritionist Pro software and used to calculate total sugar purchased from target grocery stores each week. For this analysis, the weekly values were aggregated, such that the least squares means reported herein represent average sugar (grams) purchased across all 5 weeks, in the context of the repeated measures ANOVA model.
Time Frame: Weeks 1-5 (testing overall main effect of study group)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: grams
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 21 | 21 | 23
grams | 1271.2 (905.47) | 1110.85 (902.90) | 1035.17 (907.99)

9. Primary Outcome: Change in Sugars Purchased
Description: Receipt data will be entered into Nutritionist Pro and will be used to calculate changes in sugars purchased from target grocery stores.
Time Frame: Baseline (week 1), intervention (weeks 2-4), and post-test (week 5)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
grams | -138.31 (265.25) | -374.92 (264.84) | -308.32 (249.56)

10. Primary Outcome: Nutritional Quality of Purchases
Description: Nutritional quality of grocery purchases was created using indicators adapted from Fung 2008: fruit, vegetables, nuts/legumes, whole grains, low-fat dairy, sodium, red/processed meat, carbohydrates. Quintiles were calculated for each, using the number of items from a food group or sodium [mg] and carbohydrates [g] purchased that week. Resulting scores from 1-5 indicate whether participants were lower or higher on each indicator (red meat, sodium, carbohydrates reverse scored). The 8 scores were summed for a total nutritional quality score ranging from 8 to 40 (40=highest nutritional quality).
Time Frame: At post-test (week 5)
Population: Represents those with receipt data at post-test (week 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
units on a scale | 20.89 (4.37) | 20.42 (3.22) | 21.55 (3.02)

11. Primary Outcome: Nutritional Quality of Purchases
Description: as for outcome 10
Time Frame: Weeks 1-5 (testing overall main effect of study group)
Population: All randomized participants analyzed in repeated measures ANOVA. Results reflect the average nutritional quality of purchases across all 5 study weeks (week 1-5) by group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 21 | 21 | 23
units on a scale | 20.95 (2.55) | 21.43 (2.54) | 23.86 (2.56)

12. Primary Outcome: Change in Nutritional Quality of Purchases
Description: as for outcome 10
Time Frame: Baseline (week 1), intervention (weeks 2-4), and post-test (week 5)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
units on a scale | -1.47 (1.13) | -2.04 (1.13) | -1.39 (1.06)

13. Secondary Outcome: Dollars Spent
Description: Total dollars spent at the target grocery stores from submitted receipts
Time Frame: At post-test (week 5)
Population: Sample sizes reflect those providing receipt data in week 5.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
dollars | 84.71 (47.05) | 88.79 (61.52) | 72.59 (42.19)

14. Secondary Outcome: Dollars Spent
Description: Total dollars spent at the target grocery stores from submitted receipts
Time Frame: Weeks 1-5 (testing overall main effect of study group)
Population: Results reflect the least squares means in each group across all 5 weeks of receipt data collection in the context of the repeated measures ANOVA model. In other words, results below can be thought of as average dollars spent by each study group over the course of the 5-week study.
Measure: Least Squares Mean (Standard Error); unit: dollars
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 21 | 21 | 23
dollars | 88.93 (10.76) | 87.64 (10.74) | 80.69 (10.31)

15. Secondary Outcome: Change in Dollars Spent
Description: Changes in total dollars spent at the target grocery stores from submitted receipts
Time Frame: Baseline (week 1), intervention (weeks 2-4), and post-test (week 5)
Population: The results below represent the change in dollars spent when purchasing groceries from target stores from week 1 to week 5 in each study group.
Measure: Least Squares Mean (Standard Error); unit: dollars
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 19 | 19 | 22
dollars | -7.20 (11.78) | -8.65 (11.76) | -24.72 (11.09)

16. Secondary Outcome: Nutritional Quality of Foods Consumed
Description: Nutritional quality of grocery purchases was created from food frequency questionnaire data using indicators adapted from Fung 2008: fruit, vegetables, nuts/legumes, whole grains, low-fat dairy, sodium, red/processed meat, carbohydrates. Quintiles were calculated for each, using reports of the frequency that the food group or nutrient of interest was consumed over the past month. Resulting scores from 1-5 indicate whether participants were lower or higher on each indicator (red meat, sodium, carbohydrates reverse scored). The 8 scores were summed for a total nutritional quality score ranging from 8 to 40 (40=highest nutritional quality).
Time Frame: At post-test (week 5)
Population: The total sample size of participants with usable food frequency questionnaire is 55 out of the 65 randomized participants. The outcome data provided is from the final intake model; least squares means are provided for each study group after adjusting for two covariates that warranted inclusion in the model, participant gender and income.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
Number analyzed (Participants) | 18 | 18 | 19
units on a scale | 20.99 (1.32) | 21.13 (1.35) | 22.00 (1.33)

ADVERSE EVENTS:
Time Frame: We monitored for adverse events for each participant from their baseline assessment through study completion, an average of 5 weeks.
Arm/Group | Group 1 - Control | Group 2 - Online | Group 3 - Default
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT04051008/Prot_SAP_000.pdf